CLINICAL TRIAL: NCT02854150
Title: Improving Genetic Counseling for Patients With Spina Bifida Using Next Generation Sequencing
Acronym: EXOSPINA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC14_9736
Record Dates: First submitted 2016-07-26; First posted 2016-08-03 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Spina Bifida
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: characterization of variants in new genes using high throughput sequencing either on a panel of targeted genes or on exome in families.

SUMMARY:
The main objective is to improve genetic counseling in patients with Spina Bifida, by the characterization of variants in new genes using high throughput sequencing either on a panel of targeted genes or on exome in families.

ELIGIBILITY:
Inclusion Criteria:

* Spina Bifida patients (without age restriction), attending the genetic consultation at the National Reference Centre for Spina Bifida. These patients gave their written agreement for studying genes which could be involved in Spina Bifida.

Exclusion Criteria:

* Patients who refused to give their authorization to perform the sequencing of genes involved in Spina Bifida on their DNA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Spina Bifida patients (without age restriction), attending the genetic consultation at the National Reference Centre for Spina Bifida
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
absence or low frequency (<1%) in public databases (dbSNP, Hapmap, 1000Genome) | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier universitaire de RENNES, Rennes, France